CLINICAL TRIAL: NCT03599414
Title: CASPA (CArdiac Sarcoidosis in PApworth): Improving the Diagnosis of Cardiac Disease in Patients With Pulmonary Sarcoidosis
Brief Title: CASPA: CArdiac Sarcoidosis in PApworth
Acronym: CASPA
Status: Completed | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: P02262
Record Dates: First submitted 2018-06-05; First posted 2018-07-26 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Interstitial Lung Disease; Pulmonary Sarcoidosis; Cardiac Sarcoidosis
Keywords: sarcoidosis; cardiac; MRI; Echocardiography; pulmonary; cytokine
MeSH Terms: conditions — Lung Diseases, Interstitial; Sarcoidosis, Pulmonary; Sarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sarcoidosis is a disease of unknown cause which affects adults of all ethnic backgrounds. Clumps of tissue called granulomas develop primarily in the lungs, but can damage other organs, especially the heart. Anecdotal evidence from autopsy studies suggests the heart is affected in up to 68% of patients, but there is much uncertainty about this figure.

If undetected and untreated, it can lead to serious complications or even sudden death. The current recommendation is to perform heart tracings (ECG s) on all patients, but this detects fewer than half of those with heart involvement.

Blood markers traditionally used to diagnose heart disease are unreliable, meaning there is no simple blood test in use.

The investigators propose a study with three aims. Firstly, identify the true prevalence of heart disease by performing Magnetic Resonance Imaging (MRI) scans on a group of patients with newly diagnosed lung sarcoidosis. Those found to have heart disease will have specialist (but routine) electrical heart tests. Secondly, (and perhaps the most immediate and clinically relevant) to identify the best method of diagnosing heart involvement using a combination of three simple tests: advanced ECG, 24-hour continuous ECG and a new type of computerised ultrasound scan. Thirdly, to identify proteins in the blood that could be used to develop a simple blood test for heart involvement in patients with lung sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

* Newly referred adult patients with pulmonary sarcoidosis and diagnosis made at multidisciplinary meeting as per current joint BTS/ATS guidance
* Patient may be on ≤10mg prednisolone at time of recruitment (if already started at another site prior to referral).
* Able to give informed consent and able to comply with protocol
* ≥>18 yrs

Exclusion Criteria:

* History of other cardiac disease (e.g. coronary artery disease)cardiac surgery or previous myocardial infarction (MI)
* Inability to give informed consent
* <18 yrs
* Patient may be on >10mg prednisolone at time of recruitment (if already started at another site prior to referral).
* On non-steroidal medication including methotrexate
* Pregnancy
* Alcoholism
* Illicit drug abuse

Exclusion criteria for MRI:

* Cardiac pacemakers
* Surgical clips in the head (particularly aneurysm clips)
* Electronic inner ear implants (bionic ears)
* Ocular metal fragments • Electronic stimulators • Implanted pumps
* Severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of pulmonary sarcoidosis
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
The prevalence of cardiac sarcoidosis in patients with pulmonary sarcoidosis | on Day 1
  The prevalence of cardiac sarcoidosis in patients with pulmonary sarcoidosis

SECONDARY OUTCOMES:
Cytokine and Proteomic profiling | after 1 year
  Completion of cytokine and proteomic profiling of patients with pulmonary sarcoidosis
Diagnosis of cardiac sarcoidosis | on Day 1
  Diagnosis of cardiac sarcoidosis by combining signal averaged ECG, speckle tracking echocardiography and 24 hour holter monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Muhunthan Thillai, Principal Investigator — Royal Papworth Hospital
Locations (1):
- Royal Papworth Hospital, Papworth Everard, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No